CLINICAL TRIAL: NCT06860841
Title: Effects of D-Chiro-Inositol Combined with Metformin on Insulin Resistance in People with Overweight or Obesity and Type 2 Diabetes Mellitus: a Placebo-controlled Randomized Double-Blind Crossover Trial
Brief Title: Effects of D-Chiro-Inositol Combined with Metformin on Insulin Resistance in People with Overweight or Obesity and T2DM
Acronym: DIACHIRO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Silvia Manfrini, Prof., MD, Campus Bio-Medico University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: The DIACHIRO Study
Record Dates: First submitted 2025-02-21; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Overweight and Obese Adults
Keywords: D-Chiro-Inositol; Type 2 Diabetes Mellitus; Insulin Resistance; Metformin; Glycemic Variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention/Treatment (Experimental): D-Chiro-Inositol in combination with metformin
  Interventions: Drug: D-Chiro-Inositol Combined with Metformin
- Active Comparator Intervention/Treatment (Active Comparator): Placebo in combination with metformin
  Interventions: Drug: Placebo in combination with metformin

INTERVENTIONS:
Drug: D-Chiro-Inositol Combined with Metformin — D-chiro-Inositol will be administered for 14 days,1 cp after lunch and 1 cp after dinner in addition to preexisting metformin therapy
  Arms: Experimental Intervention/Treatment
Drug: Placebo in combination with metformin — placebo will be administerd for 14 days, 1 cp after lunch and 1 cp after dinner in addition to pre-existing metformin therapy
  Arms: Active Comparator Intervention/Treatment

SUMMARY:
This study evaluates the efficacy of D-Chiro-Inositol (DCI) as an add-on therapy to metformin in improving insulin resistance, measured by the HOMA index, in people with overweight or obesity and type 2 diabetes mellitus (T2DM). Secondary outcomes include glycemic variability, indirect calorimetry, respiratory quotient, and other metabolic parameters.

DETAILED DESCRIPTION:
The DIACHIRO trial is a randomized, double-blind, crossover clinical trial assessing the impact of DCI combined with metformin versus metformin plus placebo on insulin resistance in people with overweight or obesity and T2DM. The primary outcome is the change in the HOMA index. Secondary outcomes include glycemic variability parameters (e.g., time in range), oxidative stress markers, indirect calorimetry, respiratory quotient, and HbA1c levels. Participants are monitored using Flash Glucose Monitoring (FGM) systems.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes mellitus.
2. Age between 18-75 years.
3. BMI ≥25 kg/m².
4. HbA1c < 9%.
5. Stable dose of metformin for at least three months prior to enrollment.

Exclusion Criteria:

1. Use of antidiabetic drugs other than metformin within three months prior to enrollment.
2. History of ketoacidosis or severe hypoglycemia within six months prior to enrollment.
3. Significant renal or hepatic impairment (eGFR <60 mL/min/1.73 m²; ALT/AST >2× ULN).
4. Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in the HOMA index | at the end of treatment phase (two weeks)
  fasting glucose and insulin will be measured

SECONDARY OUTCOMES:
Time in Range in % | at the end of treatment (two weeks)
  Time in range in % (time spent with a glucose level between 70-180 mg/dL expressed in %)
Changes in oxidative stress markers | at the end of treatment (two weeks)
  D-ROM PAT
Indirect calorimetry measurements | at the end of treatment (two weeks)
  Indirect calorimetry measurements
Respiratory quotient measurements. | at the end of treatment (two weeks)
  Respiratory quotient measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No